CLINICAL TRIAL: NCT03072875
Title: CAMS Relational Agent System for Suicide Prevention
Brief Title: CAMS-RAS: for Suicide Prevention
Acronym: CAMS-RAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Evidence-Based Practice Institute, Seattle, WA (Industry)
Collaborators: The Catholic University of America (Other); University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R43MH108222-01A1 (NIH)
Record Dates: First submitted 2017-02-23; First posted 2017-03-07 (Actual); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Suicide
Keywords: Suicidality; Collaborative Assessment and Management of Suicidality; Technology; Suicide Prevention; Suicide Intervention
MeSH Terms: conditions — Suicide; Suicidal Ideation; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAMS-RAS (Experimental): In this single-arm study design, all enrolled patient participants are asked to provide feedback on the CAMS-RAS prototype as it is developed for this study. Feedback will be gathered via survey measure and interview.
  Interventions: Device: CAMS-RAS

INTERVENTIONS:
Device: CAMS-RAS

SUMMARY:
This Phase I feasibility study endeavors to create a prototype of a tool to determine its feasibility with suicidal patients in emergency departments (EDs). This is not a clinical trial. The overarching goal of this research is to create a tool that could reduce suicide rates, increase delivery of efficacious suicide interventions, and decrease overall costs associated with suicidal behaviors. SBIR Phase I project aims include: (1) creating an advisory board to guide the development of CAMS-RAS; (2) iteratively design and develop relational agent ("Dr. Dave") modeled after the gestures, expressions, and mannerisms of CAMS treatment developer, David Jobes, PhD; and (3) conduct feasibility tests to determine whether CAMS-RAS is acceptable, easy to use, and liked by target end-users: acutely suicidal patients admitted to hospital EDs, psychiatric inpatient units, and medical floors for treatment of injuries sustained during a suicide attempt; hospital medical personnel, administrators, and other stakeholders including peer advocates; and outpatient suicidal patients, clinicians and administrators.

ELIGIBILITY:
Patient Inclusion Criteria:

* English fluency
* 18 years or older
* receiving clinical care in a hospital or outpatient clinic for suicidality
* Suicidal patients currently admitted to EDs, psychiatric inpatient units, and medical floors, or patient with past (last 6 months) suicidality receiving outpatient treatment

Patient Exclusion Criteria:

* Acutely psychotic
* severely agitated (as determined by care team)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2017-12-17 (Actual); Study Completion 2017-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda Dimeff, PhD, Principal Investigator — Evidence-Based Practice Institute
Locations (1):
- Evidence-Based Practice Institute, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
Requests for use of data will be considered on a case-by-case basis. Interested researchers may send data requests to research@ebpi.org.

RESULTS

PARTICIPANT FLOW:
Groups:
- CAMS-RAS: In this single-arm study design, all enrolled patient and non-patient participants are asked to provide feedback on the CAMS-RAS prototype as it is developed for this study. Feedback will be gathered via survey measure and interview.
  CAMS-RAS
Period: Overall Study
Arm/Group | CAMS-RAS
Started | 26
Completed | 25
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | CAMS-RAS
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Age collected from 24 patient participants only (2 unknown)
  Years
    number analyzed (Participants) | 24
    (all) | 39.38 (12.76)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 6
  Female | 16
  Other | 1
  Unknown | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 3
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Usability Satisfaction and Acceptability Questionnaire (USAQ)
Description: A brief face-valid, self-report measure that the PI derived from the System Usability Scale and has been successfully used in previous studies. Items are rated on a 5-point Likert Scale (1=poor; 3=good; 5=excellent). Includes open-ended questions to better understand what was most and least helpful with respect to each category and also measures users' acceptance.
Time Frame: up to one day
Population: Suicidal ED Patients only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAMS-RAS
Number analyzed (Participants) | 6
units on a scale | 4.5 (0.41)
Statistical Analysis 1: Comparison: CAMS-RAS; Test type: Other — Descriptive statistic; Quantitative data (descriptive statistic) from the USAQ were used to determine feasibility. Specifically, we established an a priori mean score of 3.5 or greater on the USAQ to determine feasibility

2. Primary Outcome: Number of ED Patient Participants Who Completed Semi-Structured Interview
Description: A semi-structured interview was conducted following use of the CAMS-RAS tool to assess users' likes, dislikes, and other preferences. Questions included: "What were your experiences in using 'Dr. Dave' and the CAMS-RAS system?" and "What suggestions would you have for improvement?" All subjects indicated that they found the tool helpful to them. They described the tool using adjectives similar to those used to describe "Nurse Louise" - a "discharge nurse" avatar on which the investigator's avatar was based: "He's kind and asks me really practical, helpful questions"; "He speaks to me directly in a compassionate way"; and "He is kind and invested".
Time Frame: After interacting with the technology (length: approximately 1 hour), subjects were then asked to complete the semi-structured interview conducted by the research assistant. On average, the interview lasted approximately 15 minutes.
Population: The qualitative information from the semi-structured interviews tells us subjects' general opinions and preferences concerning the avatar.
Measure: Count of Participants; unit: Participants
Groups:
- CAMS-RAS: In this single-arm study design, all enrolled patient participants are asked to provide feedback on the CAMS-RAS prototype as it is developed for this study. Feedback will be gathered via survey measure and interview.
  CAMS-RAS
Arm/Group | CAMS-RAS
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | CAMS-RAS
All-Cause Mortality (participants affected / at risk) | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/26

LIMITATIONS AND CAVEATS:
This SBIR Phase I Feasibility Study endeavored to create a prototype of a tool to determine its feasibility with suicidal patients in emergency departments. This is not a clinical trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT03072875/Prot_SAP_000.pdf